CLINICAL TRIAL: NCT06302985
Title: Application of Atomized Inhalation ICG in Thoracoscopic Surgery for Pulmonary Sequestration in Children: a Multicentre Prospective Study
Brief Title: Atomized Inhalation ICG for Treatment of Congenital Lung Malformations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiexiong Feng (Other)
Responsible Party: Sponsor-Investigator, Jiexiong Feng, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICG-CLMs
Record Dates: First submitted 2024-02-21; First posted 2024-03-12 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Sequestration; Congenital Pulmonary Airway Malformation; Indocyanine Green; Thoracoscopic Surgery; Children
MeSH Terms: conditions — Bronchopulmonary Sequestration; Cystic Adenomatoid Malformation of Lung, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICG for CLMs (Experimental): Preoperative preparation ICG solution dissolved in 5ml of normal saline (dose 0.5mg/kg) was inhaled 30 minutes before surgery.
  Operation method After entering the chest cavity, the fluorescence endoscope was switched to the fluorescence display mode, and the fluorescence-stained normal lung tissue and non-stained lesion tissue could be clearly displayed through the display screen, and the external boundary of the lesion was marked with an electric hook. The mediastinal pleura and pulmonary pleura were opened along the boundary of the lesion, and the lung tissue was split along the gap between the lesion and the lung tissue with an electric coagulation hook and an ultrasonic knife, and the lesion arteries and bronchi were freed. Smaller blood vessels could be cut by Ligasure or ultrasonic knife directly, and thicker blood vessels and bronchi should be cut by Hemolock until the lesion resection was completed.
  Interventions: Procedure: atomized inhalation ICG before thoracoscope pneumonectomy

INTERVENTIONS:
Procedure: atomized inhalation ICG before thoracoscope pneumonectomy — Preoperative preparation ICG solution dissolved in 5ml of normal saline (dose 0.5mg/kg) was inhaled 30 minutes before surgery.
  Operation method After entering the chest cavity, the fluorescence endoscope was switched to the fluorescence display mode, and the fluorescence-stained normal lung tissue and non-stained lesion tissue could be clearly displayed through the display screen, and the external boundary of the lesion was marked with an electric hook. The mediastinal pleura and pulmonary pleura were opened along the boundary of the lesion, and the lung tissue was split along the gap between the lesion and the lung tissue with an electric coagulation hook and an ultrasonic knife, and the lesion arteries and bronchi were freed.

SUMMARY:
To investigate the safety and effectiveness of preoperative aerosol inhalation ICG solution for thoracoscopic accurate resection of congenital lung malformations in children.

DETAILED DESCRIPTION:
Preoperative preparation Preoperative evaluation of pulmonary ventilation function and enhanced CT examination of the lungs were performed. Respiratory symptoms should be improved first in case of complicated respiratory infection. ICG solution dissolved in 5ml of normal saline (dose 0.5mg/kg) was inhaled 30 minutes before surgery.

Operation method Intraoperative fluorescence thoracoscopic imaging was used, and focal resection was performed. All patients were placed in lateral decubitus position under general anesthesia, and single lung ventilation was selected. A low flow rate (1-2 L/min) and low CO2 pressure (4-5 mmHg) were maintained in the thorax to establish an artificial pneumothorax. The observation hole is in the 7th or 8th intercostal space of the midaxillary line, and the two operating holes are in the 4th or 5th intercostal space of the anterior axillary line and the 8th or 9th intercostal space of the posterior axillary line, respectively. 30 degrees 10 mm fluorescence thoracoscope. After entering the chest cavity, the fluorescence endoscope was switched to the fluorescence display mode, and the fluorescence-stained normal lung tissue and non-stained lesion tissue could be clearly displayed through the display screen, and the external boundary of the lesion was marked with an electric hook. The mediastinal pleura and pulmonary pleura were opened along the boundary of the lesion, and the lung tissue was split along the gap between the lesion and the lung tissue with an electric coagulation hook and an ultrasonic knife, and the lesion arteries and bronchi were freed. Smaller blood vessels could be cut by Ligasure or ultrasonic knife directly, and thicker blood vessels and bronchi should be cut by Hemolock until the lesion resection was completed. After the lesion was removed, the chest was rinsed with warm normal saline, and the lung tissue section was carefully examined to confirm that there was no active bleeding and air leakage, and the lung was well dilated. The intercostal nerve was blocked under thoracoscopic vision. Finally, the thoracic closed drainage tube was placed in the midaxillary line puncture hole and the incision was closed.

Post-operation follow-up All patients undergo outpatient follow-up 3-6 months after surgery, including pulmonary CT and pulmonary ventilation function measurements, and comparison of VT (tidal volume), Ti/Te suction/exhalation time ratio, TPTEF/TE (peak time ratio) and VPEF/VE (peak volume ratio) before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* children with congenital lung malformations diagnosed by CT or MRI scan

Exclusion Criteria:

* 1. ages <3 months and >14 years 2. complicated other life-threatening disease; 3. complicated severely pulmonary infection

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
rate residual | 3 months
  Residual lesions can usually only be found in postoperative radiology scan

SECONDARY OUTCOMES:
peak volume ratio | 3 months
  Pulmonary function review ventilator-function indicators of peak volume ratio
length of hospital stay | up to 14 days
  length of hospital stay
peak time ratio | 3 months
  Pulmonary function review ventilator-function indicators of peak time ratio

CONTACTS AND LOCATIONS:
Overall Officials: Tianqi Zhu, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China